CLINICAL TRIAL: NCT07159724
Title: Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the Usefulness, Satisfaction, and Ease of Use Questionnaire (USE) in Individuals With Back and Neck Pain
Brief Title: Turkish Version of the Usefulness, Satisfaction, and Ease of Use Questionnaire (USE): Reliability and Validity
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ABDURAHİM ASLIYÜCE, Research Assisstant, Hacettepe University
Other Study IDs: FTREK24/39
Record Dates: First submitted 2025-08-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Neck Pain; Low Back Pain; Biomedical Technology; Validation
Keywords: Musculoskeletal Pain; validaiton; medical device; evaluation
MeSH Terms: conditions — Neck Pain; Low Back Pain; Musculoskeletal Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with low back and neck pain: Participants will be adults aged 18-65 years who have experienced low back or neck pain for at least 3 months and have undergone rehabilitation including at least one biomedical device (e.g., Back Up, Mollii Suit, Compex, or TENS). Eligible individuals must be literate and willing to provide informed consent. Exclusion criteria include malignancy, pregnancy, neurological or systemic disease causing functional loss, recent surgery within the last 6 months, acute infection, unhealed fracture, or withdrawal of consent.
  Interventions: Device: back up, mollii-suit, compex, tens

INTERVENTIONS:
Device: back up, mollii-suit, compex, tens — In order to be included in this study, individuals must have undergone at least one session of treatment with a biomedical device.
  In the validity and reliability study of the Turkish version of the questionnaire, permission was first obtained from the questionnaire's author via e-mail. The Usefulness, Satisfaction and Ease of Use Questionnaire (USE) was translated from English into Turkish by two independent translators: one was a physiotherapist with a doctoral degree, and the other a faculty member at Hacettepe University School of Foreign Languages. Both translators were native Turkish speakers, fluent in English, and had no personal or professional interaction with each other. They evaluated the original questionnaire in terms of meaning and grammar to produce the Turkish version of the Usefulness, Satisfaction and Ease of Use Questionnaire (USE).
  The independently translated Turkish versions of the questionnaire were then reviewed by an expert panel to reach consensus. This exp

SUMMARY:
In recent years, numerous technological products and devices have been developed in rehabilitation through advances in biomedical technology. These innovations support traditional rehabilitation services, offering more effective treatment methods and improving patients' adherence and participation. Increased compliance in treatment positively influences functional status, quality of life, and satisfaction. However, the diversity of biomedical products and the varying strength of their scientific foundations make it critical to evaluate them in terms of benefit, patient compliance, and usability. In physiotherapy and rehabilitation, objective tools for this purpose remain limited, which hinders accurate assessment of product effectiveness and the identification of improvements. Uncertainty regarding usability and ease of use may also result in inefficient utilization of resources.

Questionnaires provide cost-effective tools to capture users' opinions, reflecting strengths and weaknesses of a product without the need for measurement devices. The Usefulness, Satisfaction, and Ease of Use (USE) Questionnaire, developed by Arnold Lund in 2001, is a comprehensive 30-item scale scored on a 7-point Likert system. It evaluates usefulness, ease of use, ease of learning, and satisfaction, with items applicable across different products and services such as software, hardware, applications, or user support materials. Its multidimensional structure allows for the evaluation of usability in physiotherapy and rehabilitation technologies as well as in broader fields including robotics, social networking sites, diagnostic tools, and virtual reality.

Despite its wide use internationally, no validated Turkish version of the USE Questionnaire exists. Establishing a culturally adapted, valid, and reliable Turkish version will address this gap and provide clinicians and researchers with a standardized tool for usability assessment.

The aim of this study is to investigate the validity and reliability of the Turkish version of the USE Questionnaire.

DETAILED DESCRIPTION:
This study will be carried out at Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Spine Health Unit. Individuals who apply to the rehabilitation program and use biomedical devices will be included. Inclusion criteria are: presence of back or neck pain for at least three months, use of a supportive biomedical device in the rehabilitation program, literacy, age between 18-65 years, and voluntary participation with written informed consent. Exclusion criteria include malignancy, pregnancy, neurological or systemic disease causing functional loss, surgery within the last six months, acute infection, unhealed fracture, or withdrawal of consent at any stage.

The cross-cultural adaptation of the Usefulness, Satisfaction and Ease of Use (USE) Questionnaire will be conducted according to established guidelines. Permission has been obtained from the original author. Two bilingual translators (a physiotherapist with a PhD and a linguist from Hacettepe University School of Foreign Languages) will independently translate the questionnaire into Turkish. Their translations will be reviewed by an expert committee consisting of three health professionals and three linguists. Back-translation into English will be performed by two native English speakers. Following review and consensus, a pre-final Turkish version will be created. The pre-test phase will include 10 individuals with back or neck pain who used biomedical devices in rehabilitation. Comprehensibility, clarity, and time to complete the questionnaire will be evaluated. Items that are unclear will be revised or removed.

A total of 150-300 participants will be recruited, following the recommendation of 5-10 participants per item for validation studies. Data collection will include demographic information (age, sex, weight, height, occupation, education, diagnosis), the Turkish USE Questionnaire, Neck Disability Index, Oswestry Disability Index, Quebec User Evaluation of Satisfaction with Assistive Technology, and Numeric Pain Rating Scale. Device-related usefulness, learning, and ease of use will be evaluated using Visual Analog Scales. The USE Questionnaire will be administered twice, with a three-day interval, to assess test-retest reliability.

Statistical analyses will be performed using IBM SPSS. Construct validity will be examined using factor analysis and correlations with established scales. Internal consistency will be assessed by Cronbach's alpha coefficient, and test-retest reliability will be evaluated using intraclass correlation coefficients. These methodological steps will ensure the scientific rigor, validity, and reliability of the Turkish version of the USE Questionnaire. The adapted instrument is expected to provide a standardized and reliable tool to evaluate usability of biomedical devices and technologies in physiotherapy and rehabilitation settings, filling an important gap in the Turkish literature.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of back or neck pain lasting at least 3 months
2. Use of a supportive biomedical device in a rehabilitation program
3. Literacy
4. Age between 18 and 65
5. Willingness to participate in the study on a voluntary basis

Exclusion Criteria:

* 1. Malignant condition 2. Pregnancy 3. Loss of function due to neurological or systemic disease 4. Having undergone surgery in the last 6 months 5. Acute infection 6. Unhealed fracture 7. Withdrawal from any phase of the study 8. Light sensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with low back pain and neck pain
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Baseline (Day 1)
  It was developed by Vernon and colleagues as a neck version of the Oswestry Back Pain Scale. The Turkish version was developed by Aslan and colleagues. The Neck Disability Questionnaire consists of a total of 10 questions related to pain, personal care, concentration, work, driving, and sleeping. Each question is scored on a scale of 0 to 5. The total score is evaluated out of 50.
Usefulness, Satisfaction, and Ease of Use Questionnaire | Baseline (Day 1) and 3 days after initial assessment
  Developed by Arnold Lund in 2001, the Usefulness, Satisfaction, and Ease of Use Questionnaire (USE) is a comprehensive tool consisting of 30 items that assess various dimensions of usability. The questionnaire is scored on a 7-point Likert scale (1 = "Strongly Disagree"; 7 = "Strongly Agree") and includes a "None" option.
Oswestry Disability Index | Baseline (Day 1)
  Developed by Fairbank et al. to assess the level of functional loss in individuals with back pain. The Turkish version was developed by Yakut et al. The scale consists of 10 questions related to pain intensity, self-care, lifting and carrying, walking, sitting, standing, sleeping, degree of pain change, travel, and social life. Each question is scored on a scale of 0 to 5. The total score is evaluated out of 100.
Quebec Assistive Technology User Satisfaction Survey | Baseline (Day 1)
  The Quebec Assistive Technology User Satisfaction Evaluation (Q-YTKMD) Questionnaire is a standardized questionnaire widely used to assess the satisfaction of individuals who use various assistive devices. The Q-YTKMD Questionnaire contains 12 items that inquire about satisfaction with assistive devices (8 items) and services (4 items). The validity and reliability of the Turkish version of the Q-YTKMD Survey have been established.

SECONDARY OUTCOMES:
Evaluation of the Benefit Level of Biomedical Devices | Baseline (Day 1)
  The benefit participants derive from the biomedical device used in the rehabilitation program process will be evaluated using the Visual Analog Scale (VAS). In the literature, the VAS has been used to assess the level of benefit provided by a product or service. Participants are asked to mark the level of benefit they have received on a horizontal line 10 cm long on a plane. The scale is marked as follows: "0: not beneficial at all" and "10: very beneficial." Scoring is based on measuring the level marked by the participant on the plane with a ruler.
Assessment of the Ease of Learning Biomedical Devices | Baseline (Day 1)
  GAS will be used to assess the ease of learning related to biomedical devices used in the rehabilitation program process. Participants are asked to mark their responses on a scale from "0: not easy to learn at all" to "10: very easy to learn." Scoring is based on measuring the level marked by the participant on a ruler.
Evaluation of the Ease of Use of Biomedical Devices | Baseline (Day 1)
  GAS will be used to evaluate the ease of use of biomedical devices used in the rehabilitation program process by participants. GAS has been used in the literature to evaluate the ease of use of a product or service . Participants are asked to mark their response on a scale from "0: not easy to use at all" to "10: very easy to use." The scoring is based on measuring the level marked by the participant on a ruler.
Pain Severity Assessment | Baseline (Day 1)
  Participants' pain intensity will be assessed using the Numerical Pain Scale (NAS). The NAS is a unidimensional measure that uses 11 numbers (ranging from 0 to 10) to measure pain intensity. The patient is asked to rate their pain on the scale, with 0 indicating no pain and 10 indicating the worst (unbearable) pain.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, PT, PhD, Principal Investigator — Hacettepe University, Faculty of Physical Therapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: Undecided